CLINICAL TRIAL: NCT06901505
Title: A Randomized, Open-Label, Active-Controlled Study Evaluating the Efficacy of Three Times Weekly Vadadustat Compared to Standard of Care ESA in Patients With Anemia of CKD Receiving In-Center Hemodialysis
Brief Title: To Evaluate the Efficacy of Three Times Weekly (TIW) Vadadustat Compared to Standard of Care ESA in Patients With Anemia of CKD Receiving In-Center Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0052; VOCAL (Other: Akebia Therapeutics)
Record Dates: First submitted 2025-03-27; First posted 2025-03-30 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Erythropoiesis-Stimulating Agent; Open-label; Vadadustat
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Hematinics; vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vadadustat (Experimental): Study drug will be administered three times a week.
  Interventions: Drug: Vadadustat
- Erythropoiesis-Stimulating Agent (ESA) (Active Comparator): Dose adjustments will be determined by hemoglobin (Hb) change and current dose of ESA, per ESA dosing protocol
  Interventions: Drug: Erythropoiesis-Stimulating Agent (ESA)

INTERVENTIONS:
Drug: Erythropoiesis-Stimulating Agent (ESA) — Administered by intra-venous (IV) infusion.
  Arms: Erythropoiesis-Stimulating Agent (ESA)
Drug: Vadadustat — 300mg, oral tablets
  Other Names: Vafseo; AKB-6548
  Arms: Vadadustat

SUMMARY:
This is a multi-center, randomized (1:1), open-label, active-controlled, pragmatic study of the efficacy of vadadustat administered three times a week compared to standard of care erythropoiesis-stimulating agent for the treatment of anemia in in-center hemodialysis participants with end-stage kidney disease (ESKD). A subset of sites will participate in a red blood cell (RBC) sub-study where changes in the phenotype of RBCs in response to vadadustat treatment relative to methoxy polyethylene glycol-epoetin beta treatment in DD-CKD participants with anemia will be assessed. A separate informed consent form (ICF) will be signed by these participants who opt to be in the RBC sub-study. Of the 350 participants in the main study, approximately 28 participants will also be enrolled into the RBC sub-study. The total duration of the study is approximately 35 Weeks including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥18 years of age.
* Receiving outpatient in-center hemodialysis for ESKD at least three times a week.
* Currently prescribed or meets criteria for ESA based on approved facility policy.
* Hb > 8 grams per deciliter (g/dl).
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20%.
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.
* For selected sites, individuals who opt to participate in the RBC sub-study must meet the following inclusion criteria:
* Currently prescribed or will be prescribed methoxy polyethylene glycol-epoetin beta.
* Hb <11.5 g/dL

Exclusion Criteria:

* Contraindication to receive vadadustat per United States prescribing information (USPI) as determined by the treating health care provider.
* Concomitant use of any hypoxia-inducible factor prolyl hydroxylase inhibitor(HIF-PHI).
* Known cirrhosis or active, acute liver disease.
* Unable to comply with study requirements or compliance with attending dialysis treatments as prescribed, or in the opinion of the treating physician or Investigator, not clinically stable to participate in the study.
* Pregnant at the time of consent (per participant self-report).
* Any other reason, which in the opinion of the Investigator, would make the participants unsuitable for participation in the study.
* For selected sites, individuals who opt to participate in the RBC sub-study must also not meet the following exclusion criteria:
* History of, or currently diagnosed with, any hematological disease, such as sickle cell disease, thalassemia, hemochromatosis, Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency, myelodysplastic syndromes, or any other blood disorder that could interfere with the study outcomes.
* Participants will receive a blood transfusion within 3 months prior to the initiation of the study.
* History of or currently diagnosed with chronic lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin (Hb) | Baseline and the mean of Week 20 to 24

SECONDARY OUTCOMES:
Number of participants reporting treatment-emergent serious adverse events (TESAEs) | Up to 29 Weeks
Proportion of participants with mean Hb levels within target range | Week 16 to Week 24
Proportion of participants receiving RBC transfusions | Up to 29 Weeks

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - DaVita Research Site, Montgomery, Alabama
  - DaVita Research Site, Hartford, Connecticut
  - DaVita Research Site, Middlebury, Connecticut
  - DaVita Research Site, Columbus, Georgia
  - DaVita Research Site #1, Minneapolis, Minnesota
  - DaVita Research Site, Minneapolis, Minnesota
  - DaVita Research Site, Henderson, Nevada
  - DaVita Research Site, Las Vegas, Nevada
  - DaVita Research Site #1, El Paso, Texas
  - DaVita Research Site, El Paso, Texas
  - DaVita Research Site #1, Houston, Texas
  - DaVita Research Site, Houston, Texas
  - DaVita Research Site #1, San Antonio, Texas
  - DaVita Research Site #2, San Antonio, Texas
  - DaVita Research Site, San Antonio, Texas
  - DaVita Research Site, The Woodlands, Texas
  - DaVita Research Site #1, Norfolk, Virginia
  - DaVita Research Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No